CLINICAL TRIAL: NCT05146817
Title: Original Protocol of Oral Cavity Care During Long-term Mechanical Ventilation : Microbiological and Clinical Effects
Brief Title: Original Protocol of Oral Cavity Care During Long-term Mechanical Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IS-0921
Record Dates: First submitted 2021-11-24; First posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Adult Patients of Intensive Care Units on Long-term Lung Mechanical Ventilation
MeSH Terms: interventions — Dental Care Team

STUDY DESIGN:
Intervention Model Description: Comparison of 2 patients' groups to assess the efficiency of the method of ventilator-associated infections prevention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional oral care in long-term mechanical ventilation ICU patients (Active Comparator): Control group - traditional protocol of oral care ( traditional tooth brushing 1 time a day + chlorhexidine rinsing
  Interventions: Other: Oral care
- Original oral care protocol in long-term mechanical ventilation ICU patients (Experimental): Treatment group - original protocol of oral care: special device for tooth brushing 3 times a day with chlorhexidine .
  Interventions: Other: Oral care

INTERVENTIONS:
Other: Oral care — Treatment group - original protocol of oral care: special device for tooth brushing 3 times a day with chlorhexidine . Control group - traditional protocol of oral care ( traditional tooth brushing 1 time a day + chlorhexidine rinsing

SUMMARY:
This is a prospective open label randomized controlled trial of the efficacy of original oral care protocol for prevention of ventilator-associated pneumonia (VAP) and ventilator-associated tracheobronchitis (VAT)in adult patients mechanically ventilated for at least 3 days

DETAILED DESCRIPTION:
The study aims to clarify the effect of of the original method of oral cavity care in adult patients of intensive care units on long-term mechanical ventilation due to the assessment of the microbiological landscape of the oral cavity, oral plaque, upper and lower respiratory tract, the incidence of ventilator-associated pneumonia (VAP) and ventilator-associated tracheobronchitis (VAT) , depending on the traditional or original protocol of the oral cavity care. Ventilator associated pneumonia is associated with significant morbidity and mortality.Inadequate oral hygiene in intensive care units (ICUs) has been recognized as a critical issue, for it is an important risk factor for ventilator associated pneumonia (VAP). VAP is an aspiration pneumonia that occurs in mechanically ventilated patients, mostly caused by bacteria colonizing the oral cavity and dental plaque. It has been suggested that improvement of oral hygiene in ICU patients could lead to a reduced incidence of VAP. Although diverse oral care measures for ICU patients have been proposed in the literature, there is no evidence that could identify the most efficient ones. Although there are several evidence-based protocols, oral care measures are still performed inconsistently and differ greatly between individual ICUs.The influence of tooth brushing to maintain good oral health in the general population has long been standard practice. However the effect of brushing in the mechanically ventilated and intubated critically ill patients to dislodge organisms from dental plaque remains largely unclear

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 years or more;
2. Mechanical ventilation more than 24 hours;
3. Expected length of mechanical ventialtion more than 72 hours;

Exclusion Criteria:

1. Aspiration at the prehospital stage
2. Community-acquired pneumonia
3. COPD or specific lung diseases
4. Сhest Injury
5. Hemo and \or pneumothorax
6. Fat embolism
7. Lung cancer
8. Severe renal and\or hepatic impairment
9. Blood platelets less than 50 000 / μl
10. Pregnancy and the period of breastfeeding;
11. Other circumstances that the researcher considers inappropriate to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Microbial growtn | 14 days
  Oral and tracheal microbial growth/inhibition

CONTACTS AND LOCATIONS:
Locations (1):
- Federal North-West Medical Research Centre, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No